CLINICAL TRIAL: NCT04107376
Title: Inspection of the Colon Using a Retrograde Viewing Device for Detection of Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Timo Rath, Prof. Dr. Timo Rath, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Ludwig Demling Endoscopy
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Adenoma; Polyps
Keywords: retroviewing; endoscopy; adenoma detection; polyp detection
MeSH Terms: conditions — Adenoma; Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retroviewing endoscopy (RVE) (Experimental): Withdrawal in every colonic segment with SFV (standard forward view) followed by another withdrawal with the retroviewing endoscope. Allocation of patients to each arm (RVE or SFVE) is done by randomization using sealed envelopes.
  Interventions: Diagnostic Test: Retroviewing endoscopy
- standard forward viewing endoscopy (SFVE) (Active Comparator): Withdrawal in every colonic segment with SFV followed by another withdrawal with SFV. Allocation of patients to each arm (RVE or SFVE) is done by randomization using sealed envelopes.
  Interventions: Diagnostic Test: Retroviewing endoscopy

INTERVENTIONS:
Diagnostic Test: Retroviewing endoscopy — The colon is inspected with a new retroviewing endoscope

SUMMARY:
During standard colonoscopy a substantial number of colorectal polyps may be missed. Previous studies have found a 12-28% of miss rate for all polyps, a 31% for hyperplastic polyps and 6-27% for adenomas. In this study it is tested whether a retro viewing endoscope can detect more colorectal polyps in comparisson to standard forward viewing endoscopy. Further, ppolyps detected, mean adenomas per Patient and withdrawal time are recorded.

ELIGIBILITY:
Inclusion Criteria:

* screening colonoscopy
* 18 years of age

Exclusion Criteria:

* inflammatory bowel disease
* inadequate bowel preparation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 8 months
  calculation of the adenoma detection rate in each arm

SECONDARY OUTCOMES:
Polyp detection rate | 8 months
  polyp detection rate in each arm
Mean number of adenomas per patient | 8 months
  Mean number of adenomas per patient in each arm
Withdrawal time | 8 months
  Withdrawal time in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided